CLINICAL TRIAL: NCT02383966
Title: A Multicenter, Randomized, Open-label, Phase III Trial to Assess Efficacy and Safety of Cetuximab When Given in Combination With Cisplatin Plus 5 Fluorouracil Versus Cisplatin Plus 5-fluorouracil Alone for the First-line Treatment of Chinese Subjects With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase III Trial to Assess Efficacy and Safety of Cetuximab for the Treatment of Chinese Participants With Head and Neck Cancer
Acronym: CHANGE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR062202-060
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (Experimental)
  Interventions: Drug: Cetuximab; Drug: Cisplatin/Carboplatin; Drug: 5-fluorouracil
- Cisplatin/Carboplatin + 5-Flurouracil (Active Comparator)
  Interventions: Drug: Cisplatin/Carboplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Cetuximab — Participants received Cetuximab as an intravenous infusion at an initial dose of 400 milligrams per square meter (mg/m^2) on Day 1 and a subsequent dose of 250 mg/m^2 on Day 8 and Day 15 of each 21-day treatment cycle.
  Other Names: Erbitux
  Arms: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil
Drug: Cisplatin/Carboplatin — Cisplatin or Carboplatin (at an equivalent dose in case of intolerability of cisplatin) was administered at a dose of 75 mg/m^2 as an intravenous infusion on Day 1 of each 21-day treatment cycle.
Drug: 5-fluorouracil — Participants received 5-fluorouracil (FU) at a dose of 750 mg/m^2/day as a continuous intravenous infusion over 24 hours a day from Day 1 to Day 5 of each 21-day treatment cycle.
  Other Names: 5-FU

SUMMARY:
This trial aimed to assess efficacy and safety of cetuximab when given in combination with chemotherapy compared with chemotherapy alone in Chinese participants with recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN) as the first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of SCCHN
* Recurrent and/or metastatic SCCHN, not suitable for local-regional treatment
* Presence of at least 1 measurable lesion according to RECIST Version 1.1
* Signed written informed consent before any trial-related activities are carried out
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Prior systemic chemotherapy, except if given as part of multimodal treatment for locally advanced disease, that was completed within 6 months before randomization
* Surgery (excluding prior biopsy for diagnosis) or irradiation within 4 weeks before trial entry
* Previous treatment with monoclonal antibody or signal transduction inhibitors targeting epidermal growth factor receptor
* Nasopharyngeal carcinoma
* Known central nervous system metastasis and/or leptomeningeal disease
* Medical or psychological condition that would not permit the participant to complete the trial or sign informed consent
* Legal incapacity or limited legal capacity
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Research site, Darmstadt, Germany

REFERENCES:
- [Result] Guo Y, Luo Y, Zhang Q, Huang X, Li Z, Shen L, Feng J, Sun Y, Yang K, Ge M, Zhu X, Wang L, Liu Y, He X, Bai C, Xue K, Zeng Y, Chang X, Chen W, Lin T. First-line treatment with chemotherapy plus cetuximab in Chinese patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck: Efficacy and safety results of the randomised, phase III CHANGE-2 trial. Eur J Cancer. 2021 Oct;156:35-45. doi: 10.1016/j.ejca.2021.06.039. Epub 2021 Aug 18. PMID 34418665
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR062202-060
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent: 31 Jul 2015, Clinical data cut-off: 19 Jan 2018.
Groups:
- Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil: Participants received Cetuximab as an intravenous infusion at an initial dose of 400 milligrams per square meter (mg/m^2) on Day 1 and a subsequent dose of 250 mg/m^2 on Day 8 and Day 15 of each 21-day treatment cycle. Cisplatin or Carboplatin (at an equivalent dose in case of intolerability of cisplatin) was administered at a dose of 75 mg/m^2 as an intravenous infusion on Day 1 of each 21-day treatment cycle. After the administration of cisplatin or carboplatin, participants received 5-fluorouracil (5-FU) at a dose of 750 mg/m^2/day as a continuous intravenous infusion over 24 hours a day from Day 1 to Day 5 of each 21-day treatment cycle. All treatments were administered up to a maximum of 6 treatment cycles, post this participants without progressive disease (PD) continued to receive monotherapy with cetuximab until occurrence of disease progression or unacceptable toxicity.
- Cisplatin/Carboplatin + 5-Flurouracil: Participants received cisplatin or carboplatin (at an equivalent dose in case of intolerability of cisplatin) was administered at a dose of 75 mg/m^2 as an intravenous infusion on Day 1 of each 21-day treatment cycle. After the administration of cisplatin or carboplatin, participants received 5-fluorouracil (FU) at a dose of 750 mg/m^2/day as a continuous intravenous infusion over 24 hours a day from Day 1 to Day 5 of each 21-day treatment cycle. All treatments were administered up to a maximum of 6 treatment cycles.
Period: Overall Study
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Started | 164 | 79
Completed | 138 | 72
Not Completed | 26 | 7
Not completed — Ongoing at clinical cut-off date | 25 | 4
Not completed — Randomized, but not treated | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) analysis set included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil | Total
Number analyzed (Participants) | 164 | 79 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.52) | 57.0 (8.99) | 57.1 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 146 | 67 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 164 | 79 | 243
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 164 | 79 | 243
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time, as Assessed by an Independent Review Committee (IRC)
Description: PFS time was defined as the time in months from the date of randomization until first observation of PD (based on imaging as assessed by IRC), or death due to any cause when death occurs within 60 days after the last tumor assessment or randomization (whichever is later). PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on trial; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 millimeter. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Every 6 weeks starting from the date of randomization until occurrence of PD, assessed up to data-cutoff (904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
months | 5.5 [5.4 to 5.6] | 4.2 [3.0 to 5.3]
Statistical Analysis 1: Comparison: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil vs Cisplatin/Carboplatin + 5-Flurouracil; Test type: Other; Hazard Ratio (HR) = 0.566, 95% CI 2-sided [0.400 to 0.803]

2. Secondary Outcome: Progression-free Survival (PFS) Time, as Assessed by the Investigator
Description: PFS time was defined as the time in months from the date of randomization until first observation of PD (radiologically confirmed by Investigator), or death due to any cause when death occurs within 60 days after the last tumor assessment or randomization (whichever is later). PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on trial; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 millimeter. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Every 6 weeks starting from the date of randomization until occurrence of PD, assessed up to data-cutoff (904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
months | 5.5 [5.5 to 5.7] | 4.6 [2.9 to 5.5]
Statistical Analysis 1: Comparison: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil vs Cisplatin/Carboplatin + 5-Flurouracil; Test type: Other; Hazard Ratio (HR) = 0.568, 95% CI 2-sided [0.406 to 0.795]

3. Secondary Outcome: Overall Survival (OS) Time
Description: The OS time was defined as the time from randomization to the date of death. If a participant was alive at the time of analysis, survival time was censored at the last date when the participant was known to be alive. If this date was after data cut-off, participants were censored at the date of data cut-off. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from date of randomization up to data cutoff (assessed up to 904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
months | 10.2 [9.3 to 11.5] | 8.4 [6.5 to 9.9]
Statistical Analysis 1: Comparison: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil vs Cisplatin/Carboplatin + 5-Flurouracil; Test type: Other; Hazard Ratio (HR) = 0.705, 95% CI 2-sided [0.502 to 0.991]

4. Secondary Outcome: Best Overall Response Rate (ORR)
Description: The Best ORR was based on imaging and classified according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria. The BOR rate was defined as the number of participants whose BOR was either complete response (CR) or partial response (PR), relative to the number of participants belonging to the trial set of interest. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 6 weeks starting from the date of randomization until occurrence of PD, assessed up to data-cutoff (904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
percentage of participants | 50 [42.1 to 57.9] | 26.6 [17.3 to 37.7]
Statistical Analysis 1: Comparison: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil vs Cisplatin/Carboplatin + 5-Flurouracil; Test type: Other; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.52 to 5.45]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was based on imaging and classified according to RECIST Version 1.1 criteria. The DCR was defined as the number of participants whose Best Overall Response is either CR, PR or stable disease (SD), divided by the number of participants belonging to the trial set of interest multiplied by 100. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on trial.
Time Frame: Every 6 weeks starting from the date of randomization until occurrence of PD, assessed up to data-cutoff (904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
percentage of participants | 75.6 [68.3 to 82.0] | 59.5 [47.9 to 70.4]
Statistical Analysis 1: Comparison: Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil vs Cisplatin/Carboplatin + 5-Flurouracil; Test type: Other; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.15 to 3.95]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was determined for participants whose BOR was either CR or PR. It was defined as the time from the first assessment of CR or PR until the event defining PFS time. PFS time was defined as the time in months from the date of randomization until first observation of PD (based on imaging as assessed by IRC), or death due to any cause when death occurs within 60 days after the last tumor assessment or randomization (whichever is later). CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 6 weeks starting from the date of randomization until occurrence of PD, assessed up to data-cutoff (904 days)
Population: ITT analysis set included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 164 | 79
Weeks | 18.1 [13.1 to 20.3] | 13.9 [8.7 to 18.1]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), Treatment Emergent Adverse Events Leading to Death and AEs Leading to Discontinuation
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state up to 30 days after last administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Time from date of randomization up to data cutoff (assessed up to 904 days)
Population: Safety analysis set included all participants who had received at least 1 dose of any trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
Number analyzed (Participants) | 163 | 76
Participants
  TEAEs | 163 | 75
  TESAEs | 46 | 21
  TEAEs Leading to Death | 11 | 8
  AEs Leading to Discontinuation | 27 | 8

ADVERSE EVENTS:
Time Frame: Time from date of randomization up to data cutoff (assessed up to 904 days)
Description: Treatment emergent serious and non-serious adverse events are reported below.
Arm/Group | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil | Cisplatin/Carboplatin + 5-Flurouracil
All-Cause Mortality (participants affected / at risk) | 105/163 | 54/76
Serious Adverse Events (participants affected / at risk) | 46/163 | 21/76
Other Adverse Events (participants affected / at risk) | 163/163 | 73/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (N=163) | Cisplatin/Carboplatin + 5-Flurouracil (N=76)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oesophageal polyp (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Infected fistula (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 6 | 4
Oral infection (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Tracheostomy infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Acid base balance abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Venous haemorrhage (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Carboplatin + 5-Fluorouracil (N=163) | Cisplatin/Carboplatin + 5-Flurouracil (N=76)
Anaemia (Blood and lymphatic system disorders) | 73 | 36
Leukopenia (Blood and lymphatic system disorders) | 55 | 24
Neutropenia (Blood and lymphatic system disorders) | 58 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 7
Palpitations (Cardiac disorders) | 7 | 4
Abdominal distension (Gastrointestinal disorders) | 15 | 3
Abdominal pain (Gastrointestinal disorders) | 11 | 1
Constipation (Gastrointestinal disorders) | 73 | 31
Diarrhoea (Gastrointestinal disorders) | 44 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 1
Mouth ulceration (Gastrointestinal disorders) | 30 | 8
Nausea (Gastrointestinal disorders) | 93 | 51
Oral pain (Gastrointestinal disorders) | 9 | 3
Stomatitis (Gastrointestinal disorders) | 44 | 13
Vomiting (Gastrointestinal disorders) | 60 | 37
Asthenia (General disorders) | 40 | 17
Chest discomfort (General disorders) | 10 | 4
Facial pain (General disorders) | 2 | 6
Fatigue (General disorders) | 9 | 1
Pyrexia (General disorders) | 42 | 12
Lung infection (Infections and infestations) | 16 | 2
Paronychia (Infections and infestations) | 13 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 4
Malaise (General disorders) | 12 | 8
Alanine aminotransferase increased (Investigations) | 12 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 2
Blood creatinine increased (Investigations) | 4 | 4
Haemoglobin decreased (Investigations) | 14 | 5
Lymphocyte count decreased (Investigations) | 6 | 5
Neutrophil count decreased (Investigations) | 47 | 20
Platelet count decreased (Investigations) | 20 | 11
Red blood cell count decreased (Investigations) | 11 | 6
Weight decreased (Investigations) | 103 | 31
Weight increased (Investigations) | 9 | 3
White blood cell count decreased (Investigations) | 62 | 25
White blood cell count increased (Investigations) | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 67 | 34
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 32 | 9
Hypochloraemia (Metabolism and nutrition disorders) | 26 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 56 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 44 | 21
Hypoproteinaemia (Metabolism and nutrition disorders) | 12 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 3
Dizziness (Nervous system disorders) | 23 | 12
Headache (Nervous system disorders) | 10 | 5
Poor quality sleep (Nervous system disorders) | 10 | 5
Depressed mood (Psychiatric disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 16 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 21 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 35 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 0
Rash (Skin and subcutaneous tissue disorders) | 77 | 1
Hypertension (Vascular disorders) | 4 | 5
Hypotension (Vascular disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT02383966/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02383966/SAP_000.pdf